CLINICAL TRIAL: NCT02405897
Title: A Study to Evaluate the Efficacy and Safety of Fenestrated Cup Forceps Versus Fenestrated Alligator Forceps for Performing Transbronchial Lung Biopsy in Patients With Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0810
Record Dates: First submitted 2015-03-23; First posted 2015-04-01 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Sarcoidosis
Keywords: flexible bronchoscopy; transbronchial lung biopsy; forceps
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cup forceps (Experimental): 4 biopsies (transbronchial lung biopsy) with Cup forceps
  Interventions: Device: Cup forceps
- Alligator forceps (Active Comparator): 4 biopsies (transbronchial lung biopsy) with Alligator forceps
  Interventions: Device: Alligator forceps

INTERVENTIONS:
Device: Cup forceps — In patients with sarcoidosis, flexible bronchoscopy and transbronchial lung biopsy using cup forceps
  Arms: Cup forceps
Device: Alligator forceps — In patients with sarcoidosis, flexible bronchoscopy and transbronchial lung biopsy using alligator forceps
  Arms: Alligator forceps

SUMMARY:
Sarcoidosis is a systemic disease that results from granulomatous inflammation that involves multiple body organs. The diagnosis requires the presence of compatible clinicoradiological features along with histologic evidence that demonstrates non-caseating.1 Mediastinal lymph nodes and the lung parenchyma are the most commonly involved structures in sarcoidosis that can be sampled by, performing various bronchoscopic techniques. In a recent study the use of alligator forceps had a better yield in comparison to cup forceps. The investigators hypothesize that use of fenestrated alligator forceps in comparison to fenestrated cup forceps will yield larger samples, thereby improving the diagnostic yield and reducing the number of biopsy samples irrespective of the stage of sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystem disorder characterized by granulomatous inflammation involving various body organs. The diagnosis is based on presence of fulfillment of compatible clinicoradiological features and histologic evidence of non-caseating granuloma after exclusion of other known causes for granulomatous inflammation.1 As the lung and mediastinal lymph nodes are the most commonly involved structures in sarcoidosis, performing various bronchoscopic techniques like endobronchial biopsy (EBB), transbronchial biopsy (TBLB) and transbronchial needle aspiration (TBNA) are needed for tissue sampling. The diagnostic yield of TBLB in sarcoidosis in stage I and II varies from 31%2 to 69.6%.3 Transbronchial lung biopsy (TBLB) is performed with flexible bronchoscopy under the effect of local anesthesia and is the most commonly used bronchoscopic procedure to diagnose a wide array of lung diseases. It is performed as an outpatient procedure and is associated with minimal complications such as bleeding, pneumothorax and others.4 The procedure can be performed either as a blindly or under fluoroscopic guidance. The yield of TBLB varies depending upon the extent of disease, size of tissue, number of alveoli, number of biopsies, whether the sample floats or not and the size of forceps.5-12 The diagnostic yield of TBLB in sarcoidosis depends on the radiological stage and varies from 50-65% in stage I to 80 to 85% in stage II.13-15 The diagnostic yield also depends on the number of biopsy specimens (ten in stage I and 4-6 in stage II and III).9,10 In a recent study comprising of 44 patients with 176 samples, the use of alligator forceps yielded larger samples with lesser incidence of complications (major bleeding, alligator v/s cup forceps respectively, 1% v/s 5.7% and pneumothorax, 4.5 %v/s 9.1%). The investigators hypothesize that use of fenestrated alligator forceps in comparison to fenestrated cup forceps will yield larger samples, thereby improving the diagnostic yield and reducing the number of biopsy samples irrespective of the stage of sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

1. patients with a clinical diagnosis of sarcoidosis undergoing flexible bronchoscopy
2. age group of 12 to 90 years;
3. hemodynamically stable (systolic BP > 100 mm Hg without the need of vasopressors); and
4. ability to provide informed consent to participate in the study.

Exclusion Criteria:

1. hemoglobin less than 8 gm/dL;
2. platelet count of less than 80000;
3. bleeding diathesis;
4. prothrombin time or activated partial thrombin time prolongation of more than 6 seconds when compared to control;
5. baseline room air saturation less than 90%;
6. pregnancy; and,
7. failure to provide informed consent.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of fenestrated alligator versus fenestrated cup forceps for transbronchial lung biopsy (Size of the tissue) | 12 months
  Size of tissue: Size of the tissue will be visually assessed as small if it does not fill the cup, medium if it fills the cup and large if comes out of the cup
Diagnostic yield of fenestrated alligator versus fenestrated cup forceps for transbronchial lung biopsy (Size of the tissue) | 12 months
  Size of tissue in millimeters during histopathology
Diagnostic yield of fenestrated alligator versus fenestrated cup forceps for transbronchial lung biopsy (histopathology) | 12 months
  Histopathology examination and findings

SECONDARY OUTCOMES:
Complication (Occurrence of bleeding) | 12 months
  Occurrence of bleeding
Complication (Occurrence of pneumothorax) | 12 months
  Occurrence of pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Agarwal, MD, DM, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- Bronchoscopy suite, PGIMER, Chandigarh, India